CLINICAL TRIAL: NCT07317700
Title: A Randomized, Open-label, Positive-controlled, Parallel-grouped, Multicenter Phase III Clinical Trial on the Efficacy and Safety of Flonoltinib Maleate Tablets in Patients With Intermediate- or High-risk Myelofibrosis
Brief Title: A Clinical Trial of Flonoltinib Maleate for Intermediate or High-Risk Myelofibrosis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMF-03
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: MF
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Flonoltinib Maleate Tablets 75mg, taken orally, qd， Administer on an empty stomach
  Interventions: Drug: Flonoltinib 75mg
- control group (Active Comparator): he dosage of Ruxolitinib Phosphate Tablets should be administered orally according to the instructions, bid， Administer on an empty stomach
  Interventions: Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Drug: Flonoltinib 75mg — Flonoltinib 75mg，qd
  Arms: Experimental group
Drug: Ruxolitinib Phosphate — Ruxolitinib Phosphate ,control group
  Arms: control group

SUMMARY:
This trial adopts a multicenter, open label, positive drug parallel controlled clinical trial design, with a planned enrollment of approximately 105 participants in the MF trial. Successful trial participants were selected and assigned to either the experimental group or the control group in a 2:1 stratified manner, with the stratification factor being the Dynamic International Prognostic Scoring System (DIPSS) prognostic grading criteria. Continuously take the test drug/control drug until it meets the withdrawal criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-80 years old (including threshold), gender not limited;
2. Patients diagnosed with primary myelofibrosis (PMF) according to WHO criteria (2016 edition) or patients diagnosed with post polycythemia vera myelofibrosis (PPV-MF) or post thrombocytopenia myelofibrosis (PET-MF) according to IWG-MRT criteria;
3. Expected survival period greater than 24 weeks;
4. ECOG score 0-2 points;
5. Splenomegaly: Palpation of the splenic margin reaching or exceeding 5cm below the rib (distance from the intersection of the left clavicle midline and left rib margin to the farthest point of the spleen); Or due to physical reasons (such as obesity), it may not be palpable, but MRI/CT spleen evaluation during screening confirms a volume of >= 450 cm^3;
6. Within 7 days prior to randomization, the main organ functions were generally normal, meeting the following criteria: ALT and AST <= 2.5 × ULN; TBIL<=2.0×ULN； Serum creatinine <=1.5 × ULN or serum creatinine clearance rate (Ccr)>50 mL/min; INR, PT, and APTT <= 1.5 × ULN;
7. Can understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. The toxic reactions of previous anti-cancer treatments have not recovered to grade 1 or below (excluding hair loss), or have not fully recovered from previous surgeries;
2. Allergy to experimental drugs and their excipients;
3. For any significant clinical and laboratory abnormalities, the researchers believe that they affect the safety evaluators, such as: a. uncontrollable diabetes - fasting blood glucose>250 mg/dL (13.9 mmol/L), b. hypertension and cannot be reduced to the following range after treatment with two or more antihypertensive drugs (systolic blood pressure<160 mmHg, diastolic blood pressure<100 mmHg), c. peripheral neuropathy;
4. Patients with a history of congestive heart failure (NYHA grade III or above), unstable angina or myocardial infarction, cerebrovascular accidents or thromboembolism within the first 6 months of screening;
5. Individuals with impaired cardiac function (those with ejection fraction<45% detected by echocardiography, congenital ventricular arrhythmia, QTcF>450 ms on electrocardiogram (males), QTcF>470 ms on electrocardiogram (females), or those with arrhythmia requiring treatment at the time of screening);
6. Patients with congenital or acquired bleeding disorders or unstable thrombotic diseases requiring anticoagulant therapy;
7. Any active infection requiring systemic treatment (oral, intravenous, subcutaneous, intramuscular, etc.) within the first 14 days of randomization;
8. Active infection of hepatitis B virus (HBV) or hepatitis C virus (HCV), except for the following patients: a) HBV infection: patients who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and undergo peripheral blood HBV-DNA testing, with the lower limit of HBV-DNA detection value (i.e. the upper limit of normal value in the laboratory of each research center) can be enrolled; If the baseline HBsAg is positive, continuous antiviral treatment is required after enrollment, and HBV-DNA testing should be conducted every 12 weeks and at EOT visits; b) Patients who are positive for HCV serology but negative for HCV-RNA can be included in the study;
9. Patients who are positive for human immunodeficiency virus antibodies (HIV Ab) or anti Treponema pallidum antibodies (TP Ab) (Treponema pallidum antibodies positive);
10. Patients with epilepsy or those taking psychotropic or sedative drugs during screening;
11. Pregnant or lactating female patients, female/male patients with fertility who refuse to use contraceptive measures during the trial period and within 6 months after the trial ends;
12. Patients who have suffered from other malignant tumors within the past 5 years before the first administration (excluding cured carcinoma in situ and basal cell carcinoma of the skin);
13. Patients with combined swallowing difficulties;
14. Patients who participated in clinical trials of other new drugs or medical devices within the first month of randomization and took the study drug or used the study device;
15. Researchers believe that there are other factors that are not suitable for participating in the experiment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with >=35% reduction in spleen volume from baseline | Week 24

SECONDARY OUTCOMES:
Spleen response time: The time when the spleen volume is first observed to decrease by >=35% from baseline | Week 12,week 24
MPN-SAF TSS Total Symptom Score and Baseline Comparison Decrease | Week 2,week 4,week 8,week 12,week 24
  The MPN-SAF-TSS is used to assess the symptom burden of patients with myeloproliferative neoplasms. The questionnaire also reflects the quality of life of patients to a certain extent. During the diagnosis and treatment process, the MPN-10 questionnaire includes 10 sub symptoms (fatigue, early satiety, abdominal discomfort, poor activity, lack of concentration, night sweats, skin itching, bone pain, fever, and weight loss). Each item is graded from 0 (none) to 10 (heaviest), with a total score of 0-100 points. The higher the total score, the heavier the symptom burden.
Overall survival period | Week 2,week 4,week 8,week 12,week 24
  The time interval between the first use of medication and death caused by any reason

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Zhijian, Doctor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences (IHCAMS); Niu Ting, Doctor, Principal Investigator — West China Hospital; Miao Jia, Doctor, Principal Investigator — West China Hospital